CLINICAL TRIAL: NCT02919943
Title: Impact of Angiographic Coregistered Optical Coherence Tomography-diagnostics on Physicians Decision-making During Percutaneous Coronary Intervention in Patients With Advanced Coronary Artery Disease - the "OPTICO-Integration-Trial"
Brief Title: Observational Study of Angiographic Coregistered Optical Coherence Tomography in Patients Undergoing PCI
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, David Manuel Leistner, PD M.D., Charite University, Berlin, Germany
Other Study IDs: OPTICO-Integration I
Record Dates: First submitted 2016-09-27; First posted 2016-09-30 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention — OCT-guided Percutaneous Coronary Intervention.

SUMMARY:
To define and evaluate the impact of angiographic coregistered OCT on physicians decision-making through prospective data collection in PCI procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patient provides signed written informed consent before any study-specific procedure.
* Patients suffer from coronary artery disease (CAD) including at least one angiographically significant (>70% visual estimation) stenosis present in a native coronary artery with planned PCI.

Exclusion Criteria:

* Subjects with emergent PCI or in cardiogenic shock.
* Subjects with target left main (LM) lesion, with restenosis or stent thrombosis in the target vessel or with aorto-ostial lesion location within 3 mm of the aorta junction (both right and left).
* Extreme angulation (> 90°) or excessive tortuosity (> two 45° angles) proximal to or within the target lesion.
* Known renal insufficiency (examples being but not limited to estimated glomerular Filtration rate (eGFR) < 50 ml/kg/m2, serum creatinine ≥ 2.5 mg/dL or on dialysis).
* Any other medical condition that in the opinion of the investigator will interfere with patients safety or study results.
* Currently participating in another clinical study that interferes with study results.
* Pregnant or nursing subjects and those who plan pregnancy in the period up to 1 year following index procedure.
* Any condition that precludes the subject from undergoing PCI, for example subjects with heparin induced thrombocytopenia, or contrast allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective or ad hoc PCI, stable Angina, acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The primary study objective is the change in PCI strategy after pre-procedural ACR as compared to OCT imaging alone | 20 months

SECONDARY OUTCOMES:
Major adverse cardiac event (MACE)-rate (death, myocardial infarction, Re-angiography, Re-PCI and renal failure requiring dialysis), after recruitment. | 30 days, 6 months, and 12 months.
Change in PCI strategy after pre-procedural OCT imaging in comparison to conventional angiography alone. | 20 months
Longitudinal geographical miss (GM) with uncovered residual parts of "target lesion" at the proximal or distal reference segment of the stent. Detected by comparison between pre-PCI OCT with post-PCI OCT. | 20 months
Rate of side branch occlusions (%). | 20 months
Strategy changes based on post-procedural OCT and ACR Imaging. | 20 months

CONTACTS AND LOCATIONS:
Overall Officials: David M Leistner, PD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Department of Cardiology, Campus Benjamin Franklin, Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided